CLINICAL TRIAL: NCT05157399
Title: Quantification of the Effect of the OtoBand, a Non-invasive Vestibular Masker, on Objective Measures of Vertigo and Dizziness
Brief Title: Quantification of the Effect of the OtoBand on Objective Measures of Vertigo and Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otolith Labs (Industry)
Collaborators: Dizzy and Vertigo Institute of Los Angeles (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLith10302
Record Dates: First submitted 2021-11-24; First posted 2021-12-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Dizziness; Vertigo; Vestibular Migraine; Vestibular Neuritis; Labyrinthitis
Keywords: Vestibular weakness
MeSH Terms: conditions — Dizziness; Vertigo; Vestibular Neuronitis; Labyrinthitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants with vertigo and dizziness will be asked to participate in the study. Subjects that give consent will be entered into the study and three conditions (sham, therapeutic and no device) will be tested within an hour in a randomized sequence, with the OtoBand remaining in place throughout (turned off in the "no device" condition). The subjects will complete a Participant Questionnaire following the testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OtoBand Efficacy on Vertigo and Dizziness (Experimental): During the single site visit, participants will wear the Otoband, on the flat part of the right mastoid bone, about an inch behind the pinna and level with the ear canal. OtoBand will be set to 92dB or 98dB bone conduction level (Re: 1 Dyne). The participants will be fitted with the Otoband and will undergo the vestibular battery test. The investigator will record the outcome measurements.
  Interventions: Device: Otoband
- Placebo Device Efficacy on Vertigo and Dizziness (Placebo Comparator): Participants will wear the Otoband, on the flat part of the right mastoid bone, about an inch behind the pinna and level with the ear canal. OtoBand set to a bone conduction level 10dB lower than the level used in the experimental condition. Once fitted with the Otoband, participants will undergo the vestibular battery test. The investigator will record the outcome measurements.
  Interventions: Device: Placebo Device
- No Device (No Intervention): Participants will wear the OtoBand, but turned off, to collect baseline data. This will be randomized. The participants will be fitted with the Otoband and will undergo the vestibular battery test. The investigator will record the outcome measurements.

INTERVENTIONS:
Device: Otoband — Participants with Dizziness and Vertigo will wear the Otoband set at normal power (effective) during vestibular test battery and outcome measurements will be recorded by the investigator during site visit.
  Arms: OtoBand Efficacy on Vertigo and Dizziness
Device: Placebo Device — Participants with Dizziness and Vertigo will wear the placebo device set at low power during vestibular test battery and outcome measurements will be recorded by the investigator during site visit.
  Arms: Placebo Device Efficacy on Vertigo and Dizziness

SUMMARY:
Vestibular disorders are among the most common causes of disability in society and affect over 50% of the population over the age of 65 and a significant percentage of the younger population. Vestibular disorders have a dramatic impact on daily life impacting work, relationships, and even activities of daily living.The OtoBand has shown promise and might be beneficial for treating or improving the course of recovery from vestibular disorders.

This study seeks to quantify the effect of the study device, the OtoBand, on objective measures of dizziness and vertigo in patients with vestibular dysfunction.

The study will be conducted at a single-site and will be a blinded, randomized, placebo-controlled design in which participants do not know if they are receiving bone conducted stimulation 1) at a therapeutic level or 2) at a non therapeutic level.

DETAILED DESCRIPTION:
Vestibular disorders are among the most common causes of disability in society and affect over 50% of the population over the age of 65 and a significant percentage of the younger population. Vestibular disorders have a dramatic impact on daily life impacting work, relationships, and even activities of daily living. At the current time, the mainstay of therapy for many vestibular disorders is a physical therapy called vestibular rehabilitation. While usually highly effective, this therapy is time consuming and not universally effective, in part because of inconsistent subject compliance. The use of adjuvant devices to speed recovery has been studied but very few devices have proved beneficial; the few that have shown benefit only work in special populations and are large units that cost several million dollars.

In this study, the investigators will assay the efficacy of the OtoBand in participants with vertigo and dizziness. The OtoBand will be given to participants with vertigo and dizziness in patients with vestibular dysfunction. Participants will be recruited from patients who present at the Dizziness and Vertigo Institute of Los Angeles and for whom the Principal Investigators recommend a course of vestibular rehabilitation therapy. The OtoBand will be set at either a normal power (effective) or low power (lower than the power level thought to be effective, placebo device). Participants will not know if they are receiving receiving bone conducted stimulation 1) at a therapeutic level or 2) at a non therapeutic level.

This study seeks to determine if, in patients going to the Dizzy and Vertigo Institute of Los Angeles for vestibular rehabilitation therapy, objective measures of dizziness and vertigo are significantly changed by wearing the OtoBand.

Potential changes will be measured in the following tests:

* Subjective Visual Vertical (SVV),
* Sinusoidal Harmonic Acceleration (SHA), also known as rotary chair test
* Spontaneous Nystagmus

In this current protocol, three conditions (sham, therapeutic and no device) will be tested within an hour in a randomized sequence, with the OtoBand remaining in place throughout (turned off in the "no device" condition).

The primary endpoint of the study is to determine the change(s) induced by the OtoBand in objective measures of vestibular symptoms.

The secondary endpoints of the study include:

* Participant's questionnaire as to which level the participant believes they used first and second (sham setting vs therapeutic setting);
* Measure whether Migraine and Vestibulopathy patients experience higher benefits from a given power level as measured by objective tests (SVV, SHAs and spontaneous nystagmus);
* Measure whether Migraine and Vestibulopathy patients experience any benefit from the placebo setting.

ELIGIBILITY:
Inclusion Criteria:

* Vertigo that has been present for at least 90 days, constant or predictable with attacks at least twice a week.
* Classified as having vertigo from one of the following vestibulogenic vertigo conditions:

  * Migraine Associated Vertigo, aka Vestibular Migraine
  * Chronic Unilateral Vestibulopathy in one of three forms: Persistent Postural-Perceptual Dizziness (aka 3PD), Vestibular Neuritis, Labyrinthitis
* Score > 35 on Dizziness Handicap Inventory
* Willingness to cease vestibular suppressants for 24h prior to study.

Exclusion Criteria:

* Vertigo that first presented within the last 90 days
* Skull base surgery within the last 90 days
* Any skull implant (cochlear implant, bone conduction implant, DBS)
* Resolved vestibular dysfunction by the time of study appointment
* History of head injury within the last 6 months or currently suffering the effects of a head injury
* History of diagnosed untreated neuropsychiatric disorders (hypochondriasis, major depression, schizophrenia)
* Prior documented neurodegenerative disorders of hearing and balance including:

  * Multiple sclerosis
  * Vestibular schwannoma
  * History of Cerebrovascular disorders
* History of ear operation other than myringotomy (tube placement)
* Vitreous detachment of the retina (floaters) in the previous 90 days
* Presence of severe aphasia, and individuals who cannot provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Determine change in objective measures of vestibular symptoms, namely change in VOR Gain induced by the OtoBand. | Within 60 minute trial period.
  We measure the Gain of the Vestibular Ocular Reflex (VOR) associated with sinusoidal harmonic accelerations (SHAs) at multiple frequencies of rotation. The mean Gain across all frequencies will be computed for each three experimental conditions (OtoBand/sham/no device). The quantifiable outcome will be the deviation from nominal values of the Gain as a function of experimental condition.
Determine change in objective measures of vestibular symptoms, namely change in VOR Phase induced by the OtoBand. | Within 60 minute trial period.
  We measure the Phase of the Vestibular Ocular Reflex (VOR) associated with sinusoidal harmonic accelerations (SHAs) at multiple frequencies of rotation. The mean phase lag across all frequencies will be computed for each three experimental conditions (OtoBand/sham/no device). The quantifiable outcome will be the deviation from nominal values of the phase lag as a function of experimental condition.

SECONDARY OUTCOMES:
Participant's questionnaire as to which power level they believe were sham setting vs therapeutic setting | Within 60 minute trial period.
  Compare participants' estimation of which device provided the most benefits, to the improvement in VOR gain measured during sinusoidal harmonic accelerations (SHAs).
Measure whether Vestibular Migraine and Vestibulopathy patients experience higher benefits from a low vs high bone conduction levels as measured by outcomes of objective tests (SHAs and spontaneous nystagmus) | Within 60 minute trial period.
  Measure statistically significant changes in VOR gain as measured from Sinusoidal Harmonic Accelerations (SHAs) and spontaneous nystagmus, as a function of the OtoBand's power level and as a function of the participant's condition (vestibular migraine vs vestibulopathy)
Determine change in objective measures of vestibular symptoms, namely change in residual nystagmus following SHAs, as a function of experimental condition. | Within 60 minute trial period.
  Following sinusoidal harmonic accelerations (SHAs) in the rotary chair, we measure residual eye movements (nystagmus) for one minute at rest. The amplitude and frequency of these eye movements will be computed for each three experimental conditions (OtoBand/sham/no device). The quantifiable outcome will be the deviation from nominal values of the nystagmus as a function of experimental condition.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Pearce, AuD, Principal Investigator — Dizzy and Vertigo Institute of Los Angeles
Locations (1):
- Dizzy and Vertigo Institute of Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No